CLINICAL TRIAL: NCT06234033
Title: Understanding the Neural Mechanism Behind Sensory Processing Anomalies
Brief Title: Neural Mechanisms of Sensory Processing Anomalies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: North Denmark Region (Other Government)
Responsible Party: Principal Investigator, Daniel Skak Mazhari-Jensen, PhD-Fellow, Aalborg University
Other Study IDs: N-20200091
Record Dates: First submitted 2023-12-07; First posted 2024-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-01

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Sensory Processing Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder | interventions — Surveys and Questionnaires; Wechsler Scales

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Children with Autism Spectrum Disorder: Children with a confirmed diagnosis of autism spectrum disorder made by a qualified psychiatrist.
  Interventions: Behavioral: Discrimination Acuity test; Diagnostic Test: Transiently Evoked Otoacoustic Emission; Other: Questionnaires; Behavioral: Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V); Diagnostic Test: Clinical tests of ASD; Other: Electroencephalography (EEG) with auditory or vibrotactile stimuli
- Children with Attention-Deficit Hyperactivity Disorder: Children with a confirmed diagnosis of attention-deficit hyperactivity disorder made by a qualified psychiatrist.
  Interventions: Behavioral: Discrimination Acuity test; Diagnostic Test: Transiently Evoked Otoacoustic Emission; Other: Questionnaires; Behavioral: Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V); Other: Electroencephalography (EEG) with auditory or vibrotactile stimuli; Diagnostic Test: Clinical tests of ADHD
- Neurotypical children: Children without a known or presumed psychiatric diagnosis.
  Interventions: Behavioral: Discrimination Acuity test; Diagnostic Test: Transiently Evoked Otoacoustic Emission; Other: Questionnaires; Behavioral: Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V); Other: Electroencephalography (EEG) with auditory or vibrotactile stimuli

INTERVENTIONS:
Behavioral: Discrimination Acuity test — Estimating the just-noticeable difference of auditory loudness and vibrotactile displacement to fit a psychometric function for each modality with parameters: threshold, slope, sensitivity, and response criterion.
Diagnostic Test: Transiently Evoked Otoacoustic Emission — Examination of integrity of outer hair cells in the inner ear; with and without contralateral suppression.
Other: Questionnaires — Caregiver questionnaires send to parents online to acquire demographic information Autism Quotient (AQ), Child Behavior Checklist (CBCL6-16), Sensory Profile 2 (SP-2).
Behavioral: Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) — Estimates intelligence quotient
Diagnostic Test: Clinical tests of ASD — Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2)
  Groups: Children with Autism Spectrum Disorder
Other: Electroencephalography (EEG) with auditory or vibrotactile stimuli — Two paradigms will be used: an auditory frequency tagging paradigm with interspersed pitch oddballs and a classical sensory gating paradigm with either vibrotactile stimuli or auditory clicks.
Diagnostic Test: Clinical tests of ADHD — ADHD-Rating Scale (ADHD-RS)
  Groups: Children with Attention-Deficit Hyperactivity Disorder

SUMMARY:
To assess sensory processing anomalies in neurotypical children, children with autism spectrum disorder, and attention-deficit hyperactivity disorder, particularly within the vibrotactile and auditory sensory modalities.

DETAILED DESCRIPTION:
Neurodevelopmental disorders, such as attention-deficit-hyperactivity disorder (ADHD) and autism spectrum disorder (ASD), have been associated with a high prevalence of sensory processing anomalies. With the update of the diagnostic manuals International Classification of Diseases eleventh revision (ICD-11) and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V), more emphasis has been given to the sensory symptoms of both these disorders. The demand of reliable and valid quantitative measurements of sensory processing anomalies are therefore increasing as such metrics has the potential to assist clinical decision-making e.g., in (differential) diagnostics and treatment response evaluation and prediction. The present observational study focuses on auditory and tactile processing. Hearing and touch are two of the most frequency reported modalities in which individuals with ASD experience sensory anomalies. In addition, adequate auditory and tactile processing are presumed fundamental in the emergence of various social and cognitive functions such as the development of language. Elucidating the sensory symptoms by means of psychophysics, neuroimaging, and quantitative measures of peripheral sensory organs could elucidate the underlying (neuro)physiology of sensory anomalies in ASD and ADHD.

The present project aims to elucidate the physiological substrates of abnormal sensory processing by conducting a battery of tests in children with ASD, ADHD, and neurotypical children. First, a series of questionnaires will be administered to acquire a (clinical) description of the participants (Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V); Autism Quotient (AQ, child version); Childhood Behavioral Checklist (CBCL 6-16); ADHD-Ration Scale (ADHD-RS); Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2); Use of pharmacotherapy). A standardized caregiver-reported sensory profile questionnaire will serve as the primary outcome (Sensory Profile 2, Child version). Second, transiently evoked otoacoustic emissions will be measured in order to account for peripheral mechanisms of hearing as well as their contralateral suppression to measure efferent auditory system functioning. Third, a psychophysic task will be conducted for the purpose of estimating the just-noticeable difference to auditory loudness and vibrotactile displacement intensities followed by a subjective categorical loudness scale experiment. Finally, two electroencephalographic experiments will be performed: a frequency tagging paradigm with interspersed pitch oddballs and a classical sensory gating paradigm using vibrotactile stimuli and auditory clicks.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with either ADHD, ASD, or no diagnosis (typical development)
* Between 8-15 years old

Exclusion Criteria:

* Familiar history of schizophrenia and depression.
* Epilepsy, cerebral palsy, traumatic brain injury
* Musculoskeletal illnesses
* Hearing or visual impairment that cannot be corrected
* Lack of ability to cooperate
* Parents cannot read Danish

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population include three well-defined groups of subjects:
  1. Children with a diagnosis of ASD from the local Child and Adolescent Psychiatry clinic.
  2. Children with a diagnosis of ADHD from the local Child and Adolescent Psychiatry clinic.
  3. Neurotypical children without any psychiatric or neurologic diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensory Profile 2 | 8 minutes, answered within 1 month of the experimental session
  Caregiver questionnaire to assess sensory anomalies

SECONDARY OUTCOMES:
Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) | 1 hour 15 minutes, conducted within 1 year of the experimental session
  General intelligence quotient
Autism Quotient (AQ, child version) | 8 minutes, answered within 1 month of the experimental session
  Questionnaire addressing autistic traits
Childhood Behavioral Checklist (CBCL 6-16) | 15 minutes, answered within 1 month of the experimental session
  Questionnaire addressing various behaviors relevant to DSM-V
ADHD-Ration Scale (ADHD-RS) | 15 minutes, conducted within 1 year of the experimental session
  Questionnaire addressing behaviors related to severity of ADHD symptoms
Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2) | 1 hour, conducted within 1 year of the experimental session
  Questionnaire addressing behaviors related to severity of ASD symptoms
Use of pharmacotherapy | At time of experimental session
  Use of pharmacotherapy
Transiently Evoked Otoacoustic Emission (TEOAE) | 2 minutes, during experimental session
  Cochlear energy produced during the processing of a click sound using Titan (Interacoustics A/S, Denmark) measured in decibel (dB) above the noise floor (i.e., signal-to-noise ratio).
Contralateral suppression of TEOAE | 2 minutes, during experimental session
  The suppression effect on the TEOAE during binaural stimulation. Here, constant contralateral broadband pink noise is applied simultaneous to a ipsilateral TEOAE measurement. Thus, the measurement is similar to a TEOAE but here the outcome measure is the difference score (i.e., suppression effect) of with/without contralateral stimulation.
Categorical Loudness Scale | 5 minutes, during experimental session
  Identifying quiet threshold, loudness discomfort level, and a grading of sound intensities between (quiet threshold, soft, comfortable, loud, loudness discomfort level).
Auditory Loudness Discrimination Acuity | 5 minutes, during experimental session
  The just-noticeable difference (JND) from a reference tone intensity (65 decibel sound pressure level (dBSPL), 250 ms, 1000 Hz at interval one) to a test tone (amplitude increase between 0-15 dBSPL at interval two). The unit of JND is the change in dBSLP relative to the reference tone (ΔdBSLP).
Vibrotactile Displacement Discrimination Acuity | 5 minutes, during experimental session
  The just-noticeable difference (JND) from a reference displacement intensity (160 µm, 250 ms, 230 Hz at interval one) to a test tone (amplitude increase between 0-640 µm at interval two). The unit of JND is the change in µm relative to the reference displacement (Δµm).
Electroencephalography, sensory gating paradigm with auditory and vibrotactile stimulation | 30 minutes, during experimental session
  Gating/suppression of components in the event-related potential (ERP), beta-band power, and inter-trial phase coherence during stimulation.
Electroencephalography, frequency tagging with pitch oddball (two conditions) | 7 minutes, during experimental session
  Difference scores for half semi-tone oddball and four semi-tone oddball in pitch deviation.
  1. Frequency domain amplitude for the standard and oddball (1.6 and 8 Hz)
  2. Narrow-band filtered EEG amplitudes (1-17 Hz)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science and Technology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No